CLINICAL TRIAL: NCT02632032
Title: Impact of a Diabetes Camp on Glycemic Control Among Children and Adolescents Living With Type 1 Diabetes in Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Mesmin Dehayem Yefou, Consultant internist and endocrinologist, Yaounde Central Hospital, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDiC-01
Record Dates: First submitted 2015-12-04; First posted 2015-12-16 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; children; diabetes camps; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin therapy and diabetes education (Other): Children and adolescents living with type 1 diabetes already on insulin therapy received collective diabetes education during a five days camp.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Monitoring insulin therapy of campers based on their usual regimen (one of the following):
  * premixed insulin in the morning and evening,
  * premixed insulin in the morning, regular insulin in the afternoon and premixed insulin in the evening,
  * regular insulin in the morning and afternoon, and premixed insulin in the evening.
  Education of campers on different aspects of diabetes care:
  * monitoring of blood glucose
  * injection of insulin
  * adaptation of insulin doses according to blood glucose and during exercise
  * correction of hypoglycemia
  * dietary advice
  Other Names: regular, NPH and premixed insulin

SUMMARY:
Therapeutic education is central to the management of diabetes, especially in children and adolescents. Camps represent an ideal environment for education. During camps, the campers receive both theoretical and practical information intended to improve their understanding and self-management of diabetes. The metabolic impact of diabetes camp is little known among children and adolescents living with type 1 diabetes in sub-Saharan Africa. The aimed of this study was to assess the changes in glycemic control and insulin doses in a group of children and adolescents living with type 1 diabetes in Cameroon during and after camp.

DETAILED DESCRIPTION:
Participants and setting:

In this study, the investigators analyzed the data of children and adolescents living with type 1 diabetes in Cameroon who attended the diabetes camp organized in Yaoundé in July 2013 and who came back for follow up at the CDiC clinic of the Yaoundé Central Hospital, 3 and 12 months later.

The "Changing Diabetes in Children" (CDiC) project offers logistics and free medical care to children living with type 1 diabetes in Cameroon, which includes free medical consultations, insulin, syringes, a glucose meter (Accu Check Active®, Roche Diagnostics GmbH, Mannheim, Germany) glucose strips, HbA1c monitoring every 3 months, collective therapeutic education sessions every 3 months and a yearly screening for complications. All children enrolled in the project have a systematic visit every three months. During this visit, clinical and biological assessment are done, also adjustment of treatment, therapeutic education and record of data in the medical record. Many children also consult outside systematic visits to collect the material for treatment or in case of an emergency related or not with diabetes. The forms of insulin available in the project are regular insulin (Actrapid®), intermediate-acting insulin (Insulatard®) and pre-mixed insulin (Mixtard 30®). HbA1c is assessed by the in2it™ point-of-care system (Bio-Rad Laboratories, Deeside, UK).

The CDiC program organizes a 5-day camp for about 50 children twice yearly. Participants are selected by the health care personnel who follow them, based on the availability of places and on the proximity to their homes. Children of less than 6 years old, those with an acute disease and those with incomplete recovery from a previous illness are not allowed to camp.

Camp organization:

A written informed consent was obtained from parents or guardians before inclusion and a medical insurance was contracted for campers and the camp staff. The camp staff was made of a pediatric endocrinologist, an adult endocrinologist, 3 general physicians, 4 nurses, a dietician and a sport coach. The leisure program during the camp included education workshops, games, sporting activities, a visit to an animal reserve and a dinner in a restaurant in town. Meals offered to the children attending the camp were prepared following the instructions of the dietician.

Treatment protocols and insulin doses of each camper were maintained upon arrival. However, during the camp and before every meal, the dose of insulin to be injected was analyzed and eventually modified by the physician based on the results of self-monitoring of blood glucose, the quantity of carbohydrates to be ingested, and the level of physical activity to be performed. Notwithstanding, the treatment protocols could still be modified for some camper who were poorly controlled.

At the end of camp, a prescription was done for every campers and an adjustment of doses was made based on capillary glucose. Capillary glucose was measured six times a day (Before and 2 hours after the 3 main daily meals), and as needed (Before and after an intense physical activity, and in case of a symptoms suggestive of hypoglycemia). Finally, all information on each camper (injected insulin doses, capillary blood glucose, HbA1c, weight and eventual malaise) were recorded in a self-monitoring booklet by the camper always under supervision of a camp staff.

Post-camp data collection Campers were later on routinely followed at the CDiC clinic of the Yaoundé Central Hospital. Of the 46 patients who attended the camp, only 32 who came for follow up 3 and 12 months later were included in further analyses. Data on age, gender, duration of diabetes, duration of follow up in the CDiC project, weight, insulin regimen and insulin doses at the beginning, at 3 and 12 months after camp, HbA1c at the beginning, at 3 and at 12 months after camp, and the daily number hypoglycemic episodes during camp were collected. Good glycemic control was defined as HbA1c <7.5% and hypoglycemia as capillary glucose < 70mg/dl.

Data analysis Data were analyzed using the Statistical Package for Social Sciences version 12 (SPSS Inc. Chicago, IL USA). Results are presented as mean and standard deviation or median [interquartile range] for continuous variables and as count (percentage) for discrete variables. Proportions were compared by the Z test for two proportions, means by repeated measure ANOVA, paired t test or independent t test where appropriate and medians by the Wilcoxon rank sum test. Where necessary continuous variables were categorized using the median as cutoff. A p-value < 0.05 was used to characterize statistically significant results.

Ethical considerations Prior to enrolment in the CDiC project, a written informed consent form was signed by the parent or guardian authorizing the CDiC project in Cameroon to use the data obtained for research. A written informed consent was also obtained from parents or guardians before enrolment in camp. The CDiC project has also received approval from the National Ethics Committee of Cameroon (Autorisation N 271/CNE/SE/2011) to carry out research from data obtained in the project.

ELIGIBILITY:
Inclusion Criteria:

* Children living with type 1 diabetes and enrolled in the "Changing Diabetes in Children project".
* Regular follow-up at the Yaoundé Central Hospital.
* Aged between 6 and 23 years old.
* Informed consent signed by parents or guardians prior to enrollment in the CDiC project allowing investigators of the project to used data for research.
* Informed consent forms signed by parents or guardians before participation to the 2013 camp in Yaoundé.

Exclusion Criteria:

* Nonattendance of the routinely follow-up visits at the CDiC clinic Yaoundé both at 3 and 12 months after camp.

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c | Baseline to 3 months and 12 months after camp
  Comparing the mean HbA1c of campers from baseline to 3 months and 12 months after camp

SECONDARY OUTCOMES:
Changes in insulin doses | From the first day to the third day of camp, 3 months and 12 months after camp
  Comparing the mean daily insulin doses of campers from the first day to the third day of camp, and 3 months and 12 months after camp
Hypoglycemic episode per camper per day | From the first day to the third day of camp
  Comparing the mean number of hypoglycemic episode register per camper from the first day to the third day of camp
Changes in weight | Baseline to 3 months and 12 months after camp
  Comparing the mean weight of campers from baseline to 3 months and 12 months after camp

CONTACTS AND LOCATIONS:
Overall Officials: Mesmin Y Dehayem, MD, Principal Investigator — Yaounde Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dehayem MY, Takogue R, Choukem SP, Donfack OT, Katte JC, Sap S, Sobngwi E, Mbanya JC. Impact of a pioneer diabetes camp experience on glycemic control among children and adolescents living with type 1 diabetes in sub-Saharan Africa. BMC Endocr Disord. 2016 Jan 20;16:5. doi: 10.1186/s12902-016-0086-x. PMID 26791079